CLINICAL TRIAL: NCT01985880
Title: Experimental Study of Biomarker in Patient With Interstitial Cystitis/Painful Bladder
Brief Title: The Efficacy of Biomarker in Patient With Interstitial Cystitis/Painful Bladder Syndrome
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Soo Choo, M.D., Asan Medical Center
Other Study IDs: 2013-0616
Record Dates: First submitted 2013-11-10; First posted 2013-11-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Interstitial Cystitis
Keywords: Biomarkers
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — bladder biopsy, urine, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hunner's ulcer interstitial cystitis: Hunner's ulcer interstitial cystitis
- non-ulcer interstitial cystitis: non-ulcer interstitial cystitis
- Control: Control

SUMMARY:
The purpose of this study is to evaluate efficacy of biomarker in patient with interstitial cystitis/painful bladder syndrome

DETAILED DESCRIPTION:
This is a observational study

ELIGIBILITY:
Inclusion Criteria:

* 1) must have experienced bladder pain, urinary urgency and urinary frequency, for at least 6 months prior to entry into the study 2) Pain VAS ≥4 3) O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) symptom and problem ≥ 12( and pain ≥2, and nocturia ≥ 2) 4) PUF score ≥ 13 5) cystoscopic record within 2 years

Exclusion Criteria:

1. Patients who are pregnancy or, childbearing age without no contraception
2. Patients with voided volume <40 or, > 400ml
3. Patients with microscopic hematuria, (≥1+ in dipstick), If not excluded that no evidence of neoplastic tumor examination
4. Patients with urine culture showing evidence of urinary tract infection 1month prior to the study
5. Accompanied medical problem below

   * Tuberculosis in urinary system
   * Bladder cancer, urethral cancer, prostate cancer
   * Recurrent cystitis
   * anatomical disorder
6. Patients had prior surgery (eq, bladder augmentation, cystectomy
7. Patients with neurologic disorder
8. Patients with indwelling catheter or intermittent self-catheterization
9. Patients with psychologic problem

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients >20 years old with interstitial cystitis control
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
To compare of expression of the biomarker such as APF, HB-EGF, MCP-1 among the Hunner's ulcer interstitial cystitis and non-ulcer interstitial cystitis and control groups | 1month
  To compare of expression of the biomarker such as APF, HB-EGF, MCP-1 among the Hunner's ulcer interstitial cystitis and non-ulcer interstitial cystitis and control groups

SECONDARY OUTCOMES:
To compare of changes voiding parameters after bladder biopsy between Hunner' ulcer group and non-ulcer group | 1 month
  To compare of changes voiding parameters after bladder biopsy between Hunner' ulcer group and non-ulcer group
TO compare of change of scores of questionnaires such as O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q), Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF), Visual Analogue Scale (Pain) between Hunner's ulcer group and non-ulcer group | 1month
  TO compare of change of scores of questionnaires such as O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q), Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF), Visual Analogue Scale (Pain) between Hunner's ulcer group and non-ulcer group

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, M.D., Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Asan medical center Institutional review board, Seoul

IPD SHARING:
Plan to Share IPD: No